CLINICAL TRIAL: NCT01788332
Title: A Randomised Phase II Trial of Olaparib Maintenance Versus Placebo Monotherapy in Patients With Chemosensitive Advanced Non-Small Cell Lung Cancer
Brief Title: Parp Inhibitor in Advanced Non-Small Cell Lung Cancer (PIN)
Acronym: PIN
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Lisette Nixon (Other Government)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor-Investigator, Lisette Nixon, Senior Trial Manager, Velindre NHS Trust
Organization: Velindre NHS Trust (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PIN
Record Dates: First submitted 2013-02-04; First posted 2013-02-11 (Estimated); Last update posted 2018-10-26 (Actual); Status verified 2018-10

CONDITIONS: Non-small Cell Lung Cancer
Keywords: NSCLC; non-small cell; lung cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — olaparib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Olaparib (Active Comparator): 3 100mg tablets to be administered twice a day with approximately 240ml of water.
  Interventions: Drug: Olaparib
- Placebo (Placebo Comparator): 3 100mg tablets to be administered twice a day with approximately 240ml of water.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Olaparib — Olaparib is a potent inhibitor of poly (ADP-ribose) polymerase enzyme (PARP), (molecular weight 434) that is being developed as a monotherapy as well as for combination with chemotherapy and other anti-cancer agents. Olaparib can lead to tumour regression in patients with DNA repair deficient NSCLC. Olaparib may also enhance the DNA damaging effects of chemotherapy.
  Other Names: AZD2281; KU-0059436
  Arms: Olaparib
Other: Placebo — 3 100mg tablets to be administered twice a day with approximately 240ml of water
  Arms: Placebo

SUMMARY:
In 2010, more than 35,000 people died in the United Kingdom from lung cancer, the majority from non-small cell cancer (NSCLC). Chemotherapy is one of the main treatments for patients with NSCLC but those treated will still only live for an average of 9 or 10 months after diagnosis.

The purpose of this clinical trial is to find out whether or not giving a drug called Olaparib following chemotherapy will benefit patients with NSCLC who have responded to initial chemotherapy treatment by prolonging the time before the tumour regrows. Olaparib is a new, oral drug developed by AstraZeneca which may help to slow down cancer growth. The rationale for this clinical trial is that chemotherapy damages tumour cell DNA and NSCLC tumours that respond to chemotherapy are less able to repair this damage. This can be exploited by using Olaparib as it blocks an enzyme called Poly (ADP-ribose) polymerase (PARP) which is essential for DNA repair. This will prevent DNA repair and cause cancer cell death by a mechanism known as synthetic lethality. Synthetic lethality arises when a combination of mutation in two or more genes leads to cell death.

Up to 300 patients who are to receive standard chemotherapy treatment will be initially registered into the trial. Of these patients, 114 patients who have responded to chemotherapy will be randomly allocated to receive either Olaparib or an inactive dummy pill or placebo by mouth. The trial will assess whether Olaparib delays disease progression following standard chemotherapy treatment in patients. It will also show whether the side effects of adding Olaparib following standard treatment are acceptable.

DETAILED DESCRIPTION:
This is a multicentre randomised phase II trial. Patients are initially registered either before or during induction chemotherapy, their response to which will be used to determine whether they are eligible for randomisation. All patients will be asked to consent to archival tissue collection for translational analysis and to provide a translational blood sample. The second consent will precede randomisation to one of two groups of maintenance therapy (olaparib or placebo) with 1:1 randomisation if they have had an objectively measured complete or partial response following standard chemotherapy.

Randomised patients will receive olaparib or placebo until disease progression. They will be monitored by CT scan every two cycles until disease progression, where they will be managed according to local practice. Follow up will be for a maximum of 12 months from the point of randomisation or until disease progression.

All randomised patients for whom we have a baseline translational blood sample will be asked to provide a follow up blood sample upon randomisation and again at radiological progression. Registered patients with progressive disease after the initial induction chemotherapy will be asked to provide a follow-up blood sample at the end of induction chemotherapy.

ELIGIBILITY:
Inclusion Criteria - Registration (Stage 1):

* Histological diagnosis of NSCLC. Histology can be either squamous or non-squamous.
* Stage IIIB or stage IV lung cancer that is not amenable to curative therapy.
* Have had no prior systemic chemotherapy for advanced NSCLC. Previous adjuvant or neoadjuvant chemotherapy for non-advanced disease is acceptable. Prior treatment with an oral targeted therapy for e.g. EGFR/ALK or other driver- oncogene mutated lung cancer is allowed. Immunotherapy e.g. with a PD1 or PDL1 targeted agent is allowed.
* Patients who have already started their induction chemotherapy are not eligible for stage 1 of the trial
* Eligible to receive standard platinum doublet-based chemotherapy.
* Men or women, aged 18 or over and capable of giving informed consent.
* Willing to consent to provide tissue and blood for translational research.
* Informed consent prior to any study specific procedures.

Exclusion Criteria - Registration (Stage 1):

* Evidence of small cell, large cell neuroendocrine or carcinoid histology.
* Have a serious or uncontrolled medical condition that could compromise the patients' ability to adhere to the protocol.
* Have a secondary malignancy (except adequately treated non-melanomatous skin cancer, or other cancer considered cured by surgical resection or radiation). Patients who have had another malignancy in the past but have been disease free for more than 5 years are eligible.
* Previous treatment with PARP inhibitors
* Uncontrolled gastrointestinal disorders such as active diverticulitis or colitis, or any major GI resection which could have an impact on patients' ability to absorb Olaparib.
* Myelodysplastic syndrome (MDS) or acute myeloid leukaemia (AML).

Inclusion Criteria - Randomisation (Stage 2):

* Confirmed diagnosis of NSCLC (either squamous or non-squamous). Stage IIIB or stage IV that is not amenable to curative therapy.
* ECOG performance status 0-1
* Evidence of radiological response to induction chemotherapy, from the pre-treatment to baseline. This can include mixed stable/response or evidence of tumour shrinkage that does not reach the criteria of partial response according to RECIST.
* Have had no prior systemic chemotherapy for advanced NSCLC. Previous adjuvant or neoadjuvant chemotherapy for non-advanced disease is acceptable. Previous palliative radiotherapy to non-target metastases is allowed provided no more than 25% of the bone marrow volume is irradiated. Irradiated sites cannot include the sites of measurable disease unless clear tumour progression has been documented in them since the end of radiation therapy. Patients who have had adjuvant therapy and then progressed after a year of completing adjuvant therapy are eligible. Patients who have received an oral inhibitor for molecularly stratified subgroups e.g. EGFR or ALK mutated lung cancer, are allowed. Immunotherapy e.g. with a PD1 or PDL1 targeted agent is allowed.
* Adequate organ function, including the following:

  1. Adequate bone marrow reserve: White cell count ≥ 3.0 x 109/L, absolute neutrophil count (ANC) ≥ 1.5 x 109/L, platelets ≥ 100 x 109/L, haemoglobin ≥ 90g/L.
  2. Hepatic: total bilirubin ≤ 1.5 times the upper limit of normal (x ULN); alkaline phosphatase (ALP), aspartate aminotransferase (AST), or alanine aminotransferase (ALT) ≤ 2.5 x ULN. ALP, AST, and ALT ≤ 5 x ULN is acceptable if the liver has tumour involvement.
  3. Renal: calculated creatinine clearance (CrCl) ≥ 50mL/min using Cockcroft-Gault or Wright formula, serum creatinine ≤ 1.5 x institutional upper limit of normal (ULN).
  4. If blood count/morphology suggestive of MDS/AML, no features suggestive of MDS/AML on peripheral blood smear.
* Patients with reproductive potential (male or female), who are sexually active for the duration of the trial or the drug washout period, should be prepared to use two effective forms of contraception.
* Men or women, aged 18 or over.
* Willing to consent to provide tissue and blood for translational research.
* Patients must provide informed consent prior to any study specific procedures.
* There should be no more than 42 days between day 1 of the last cycle of induction chemotherapy and starting Olaparib/placebo.

Exclusion Criteria - Randomisation (Stage 2):

* Evidence of small cell, large cell neuroendocrine or carcinoid histology.
* Patients with radiological disease progression or stable disease after induction chemotherapy
* Have received treatment with an agent that has not received regulatory approval, within 30 days of study entry.
* Have had a blood transfusion within 28 days prior to commencing Olaparib or have a WBC <3 x 109/L
* Have received yellow fever vaccination in the 30 days prior to randomisation.
* Difficulty swallowing.
* Have central nervous system (CNS) metastases (unless the patient has completed successful local therapy for CNS metastases e.g. involving complete surgical removal or radical radiotherapy to a solitary CNS metastasis). A
* Concurrent administration of any other systemic antitumour therapy.
* Have a serious or uncontrolled medical condition that would compromise the patient's ability to adhere to the protocol.
* Diagnosis of a second malignancy (except adequately treated non-melanomatous skin cancer, or other cancer that is considered cured by surgical resection or radiation). Patient who had another malignancy in the past but have been disease free for more than 5 years are eligible.
* Previous treatment with PARP inhibitors.
* Uncontrolled gastrointestinal disorders such as active diverticulitis or colitis, or any major GI resection which could have an impact on patients' ability to absorb Olaparib.
* Myelodysplastic syndrome (MDS) or acute myeloid leukaemia (AML).
* Pregnant or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2014-01 (Actual); Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | 72 weeks
  To establish the anti-tumour activity of Olaparib (measured by progression free survival),we will document the time from randomisation to any disease progression and/or death, defined according to strict RECIST (Response Evaluation Criteria in Solid Tumours) v1.1. Lesions will be compared to baseline measurements to assess progression.

SECONDARY OUTCOMES:
Safety | 72 weeks
  An Independent Data Monitoring Committee will convene and assess safety when 10 and 20 patients on each arm have completed trial treatment. If the trial is deemed safe to continue then safety will be assessed again approximately every six months. Toxicity data will be assessed along with serious adverse events.
Objective response rate | 72 weeks
  This will be assessed based on radiological disease progression defined according to RECIST (Response Evaluation Criteria in Solid Tumours) v1.1.
Overall survival | 72 weeks
  This will be calculated from the time of randomisation to date of death or date last known to be alive.
Change in tumour volume reduction | 27 weeks
  Change in tumour volume reduction from randomisation to 6 months
Tolerability | 72 weeks
  This will be assessed in terms of the number of treatment reductions, delays and withdrawals.
Feasibility | 72 weeks
  Patients will complete a diary card every day to document compliance. Feasibility of use will also be assessed in terms of number of treatment reductions, delays and withdrawals.

CONTACTS AND LOCATIONS:
Overall Officials: Dean Fennell, Professor, Study Chair — University of Leicester
Locations (20):
- United Kingdom (20):
  - Blackpool Victoria Hospital, Blackpool
  - Bradford Royal Infirmary, Bradford
  - Queen's Hospital, Burton-on-Trent
  - Velindre Cancer Centre, Cardiff
  - University Hospitals Coventry and Warwickshire NHS Trust, Coventry
  - Derby Teaching Hospitals NHS Foundation Trust, Derby
  - Beatson West of Scotland Cancer Centre, Glasgow
  - Withybush General Hospital, Haverfordwest
  - Huddersfield Royal Infirmary, Huddersfield
  - University Hospitals of Morecambe Bay, Lancashire
  - St James University Hospital, Leeds
  - Leicester Royal Infirmary, Leicester
  - Charing Cross Hospital, London
  - The Christie NHS Foundation Trust, Manchester
  - The James Cook University Hospital, Middlesbrough
  - Royal Preston Hospital, Preston
  - Weston Park Hospital, Sheffield
  - University Hospitals of North Midlands, Stoke-on-Trent
  - Singleton Hospital, Swansea
  - Wrexham Maelor Hospital, Wrexham

REFERENCES:
- [Derived] Fennell DA, Porter C, Lester J, Danson S, Blackhall F, Nicolson M, Nixon L, Gardner G, White A, Griffiths G, Casbard A. Olaparib maintenance versus placebo monotherapy in patients with advanced non-small cell lung cancer (PIN): A multicentre, randomised, controlled, phase 2 trial. EClinicalMedicine. 2022 Aug 11;52:101595. doi: 10.1016/j.eclinm.2022.101595. eCollection 2022 Oct. PMID 35990583